CLINICAL TRIAL: NCT05879302
Title: Shared Decision Making for Kidney Transplant Candidates to Plan for an Organ Offer Decision
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hennepin Healthcare Research Institute (Other)
Collaborators: Mayo Clinic (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Cory Schaffhausen, Investigator, Hennepin Healthcare Research Institute
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: Pro00067603; 1R01DK134482 (NIH)
Record Dates: First submitted 2023-05-17; First posted 2023-05-30 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: End Stage Renal Disease; End-Stage Kidney Disease; Kidney Transplantation; Esrd
Keywords: Shared Decision Making; SDM; Transplantation; Organ offer; Kidney offer; KDPI
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: All study personnel involved in screening and enrollment will be masked to upcoming randomization assignments
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shared Decision Making Intervention (Experimental): Receives the Shared Decision Making Intervention
  Interventions: Behavioral: Kidney Offer Shared Decision Making
- Usual Care (No Intervention): Receives Usual Care, eg. usual patient education and counseling for kidney transplant candidates.

INTERVENTIONS:
Behavioral: Kidney Offer Shared Decision Making — The intervention consists of receiving the Donor Offer Plan (DOP), reviewing a web-based educational module about donor offers including practice offer videos, followed by a discussion about the DOP with a transplant nurse coordinator.
  Arms: Shared Decision Making Intervention

SUMMARY:
The goal of this pilot randomized trial is to learn about shared decision making in kidney transplant candidates. The aim of this proposal is to evaluate the Donor Plan Donor Choice tool to promote high-quality Shared Decision Making for providers and kidney transplant candidates at two transplant centers.

Participants will:

* Review an online education tool, Donor Plan Donor Choice.
* Discuss a Kidney Offer Plan with a transplant provider.
* Answer questions about willingness to consider different donor types.

Researchers will compare the Shared Decision Making group to usual care to generate pilot data and implementation outcomes for a larger trial.

ELIGIBILITY:
Inclusion Criteria:

* Candidate on the kidney transplant waiting list
* Greater than 3 months since listing for transplant
* 18 Years of age or older
* English-speaking

Exclusion Criteria:

* Non-English speaking
* < 18 years of age
* Patients who choose to opt out of research.
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-04-03 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Willingness to accept donor organs at risk of discard | Up to 2 months
  Willingness to accept a donor kidney offer will be measured by three items on a 5-point Likert scale anchored by "strongly agree" and "strongly disagree." Willingness to accept will be defined by answers of "agree" or "strongly agree."

SECONDARY OUTCOMES:
Knowledge | Up to 2 months
  10 Knowledge questions relating to organ offers and organ quality
Decisional Conflict | Up to 2 months
  16 Decisional Conflict questions (Ottawa scale)
Distress | Up to 2 months
  5 STOP-D (Screening Tool for Psychological Distress) questions
Shared Decision Making | Up to 2 months
  9 items of the SDMQ9 for Shared Decision Making

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Hennepin Healthcare, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No